CLINICAL TRIAL: NCT03412292
Title: A Phase I Trial of MAX-40279 Given Orally to Subjects With Acute Myelogenous Leukemia (AML)
Brief Title: MAX-40279 in Subjects With Acute Myelogenous Leukemia (AML)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Maxinovel
Record Dates: First submitted 2018-01-08; First posted 2018-01-26 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Acute Myelogenous Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAX-40279 (Experimental): MAX-40279 is provided as a capsule for oral use at 5mg, 25mg. In the dose-escalation phase, patients will be enrolled sequentially into the 5 dose levels of MAX-40279 designated in this study: 20, 40, 70, 100 and 120 mg/day (3-6 patients per cohort),bid.For each dose level, a single dose of MAX-40279 will be first administered orally followed by 1 day observation, then continuous treatment will start 4 weeks treatment (per cycle).
  After completion of the dose escalation, additional patients will be enrolled into dose expansion at the Maximum tolerated dose(MTD), up to 12 patients will be enrolled into expansion cohorts.
  Interventions: Drug: MAX-40279

INTERVENTIONS:
Drug: MAX-40279 — MAX-40279, is a multi-targeted kinase inhibitor inhibitor mainly target FLT3 and FGFR. It has a molecular weight of 496.56 Daltons, which has a formula of C24H25FN6O3S.
  MAX-40279 is yellow powder. It is insoluble in water, methanol, ethanol, 0.1 mol/L hydrochloride solution or 0.1% saline; very slightly soluble in methylene dichloride and sparingly soluble in dimethylformamide. It is stable under strong acid, strong alkali, high temperatures and exposure to light.
  MAX-40279 for clinical use is presented as a sterile yellow powder packaged in capsules at 5 mg, or 25 mg doses.
  Other Names: MAX-40279-001

SUMMARY:
This is a dose-escalation phase I trial to evaluate the safety and tolerability of MAX-40279 in subjects with acute myelogenous leukemia(AML).

DETAILED DESCRIPTION:
The class III receptor tyrosine kinase FMS-related tyrosine kinase 3 (FLT3), is mutated and activated in about 30% of adult patients with AML. The mutations involve either an internal tandem duplication (ITD) (in about 25% of AML patients) or a point mutation in the tyrosine kinase domain (TKD) (in about 7% of patients). Patients with mutations in FLT3, particularly those with ITD mutations, have a worse prognosis, with lower rate of complete remission, and lower overall survival . Thus, inhibition of activated FLT3 kinase by a pharmacologic agent is an attractive therapeutic strategy in AML.

The aberrant of fibroblast growth factor receptor (FGFR) might be a major reason fot resistance to targeted therapies, and FGFR inhibitors significantly suppress leukemia development in vivo.

MAX-40279 is a dual inhibitor of FLT3 and FGFR. Our goal is to develpe this uqiue dual inhibitor to be a more effective and wider use for AML treatment than the current known FLT3 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Ability to understand the purposes and risks of the trial and signed informed consent forms approved by the investigator's Institutional Review Board (IRB)/Independent Ethics Committee (IEC) of the trial site was obtained before the entering the trial
3. Subject has morphologically documented primary AML or AML secondary to myelodysplastic syndrome (MDS) as defined by the World Health Organization (WHO) criteria for which no established standard therapy is available
4. ECOG performance status of 0 to 2
5. Persistent chronic clinically significant nonhematological toxicities from prior treatment (including chemotherapy, kinase inhibitors, immunotherapy, experimental agents, radiation, HSCT, or surgery) must be Grade ≤ 1
6. In the absence of rapidly progressing disease clearly documented by the investigator, the interval from prior treatment to time of MAX-40279 administration will be at least 2 weeks (14 days) for prior cytotoxic agents or at least 5 half-lives for prior noncytotoxic agents, including immunosuppressive therapy post HSCT
7. Acceptable liver function defined below:

   * Total bilirubin ≤ 1.5 times upper limit of normal range (ULN)
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times ULN;
8. Acceptable renal function defined below:

   • Serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance (by the Cockcroft-Gault formula) ≥ 60 mL/min
9. Acceptable coagulation status defined below:

   * Prothrombin time < 1.3 times ULN
   * Partial thrombin time < 1.3 times ULN
10. No clinically significant abnormalities in urinalysis
11. Female participants of child bearing potential agree not to be pregnant or lactating during the study and for three months following the last dose of study drug. Both men and women of reproductive potential must agree to use a highly effective method of birth control during the study and for three months following the last dose of study drug. A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly

Exclusion Criteria:

1. Disease diagnosis of acute promyelocytic leukemia
2. Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years at the trial entry
3. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
4. Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery
5. Percutaneous coronary intervention conducted within 6 months prior to the trial entry for cardiac infarction or angina pectoris
6. Seizure disorders requiring anticonvulsant therapy
7. Taking a medication that prolongs QT interval and has a risk of Torsades de Pointes，or a history of long QT syndrome
8. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product
9. Participation in an investigational drug or device trial within 4 weeks prior to the trial entry
10. Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
11. Recent venous thrombosis (including deep vein thrombosis or pulmonary embolism within 1 year of study)
12. History of upper gastrointestinal hemorrhage, peptic ulcer disease, or bleeding diathesis
13. Subject is pregnant (positive serum beta human chorionic gonadotropin [β-HCG] test at screening) or is currently breast-feeding, their partner anticipates becoming pregnant/impregnating during the trial or within 6 months after receiving the last dose of trial treatment
14. Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial
15. Unwillingness or inability to comply with the trial protocol for any reason
16. Legal incapacity or limited legal capacity
17. Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | 8 weeks
  Incidence of treatment-related AEs
Maximum tolerated dose (MTD) | 4 weeks
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing.

SECONDARY OUTCOMES:
Tmax | First single dose(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 1 (the second dose)(pre-dose),Cycle 1 Day 15(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  Time to maximum plasma concentration
Cmax | First single dose(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 1 (the second dose)(pre-dose),Cycle 1 Day 15(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  Maximum plasma drug concentration
AUC | First single dose(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 1 (the second dose)(pre-dose),Cycle 1 Day 15(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  Area under the time-concentration curve
t1/2 | First single dose(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 1 (the second dose)(pre-dose),Cycle 1 Day 15(pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24h post-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  Observed terminal half-life
p-FLT3 Y591 | First single dose(pre-dose), Cycle 1 Day 15(pre-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  To examine the phosphorylation (activation) of either wild-type or mutated Fms-like Tyrosine Kinase-3(FLT3)
FGFR aberration | First single dose(pre-dose), Cycle 1 Day 15(pre-dose), Cycle 1 Day 28(pre-dose), Cycle 2 Day 28(pre-dose).
  To detect Fibroblast growth factor receptor(FGFR) mutation

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - St Vincent's Hospital Sydney Limited, Darlinghurst, New South Wales
  - Western NSW Local Health District, Dubbo, New South Wales
  - Monash Health, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria

IPD SHARING:
Plan to Share IPD: No